CLINICAL TRIAL: NCT00003107
Title: A Phase I Trial of Recombinant Human Interleukin-12 After High-Dose Therapy and Autologous Hematopoietic Stem Cell Support
Brief Title: Interleukin-12 in Treating Patients With Hematologic Cancers or Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Michael Robertson, MD/ Principal Investigator, Indiana University School of Medicine
Organization: Indiana University (Other)
Purpose: Treatment
Other Study IDs: 9708-05; T97-0027; IUMC-9708-05; NCI-T97-0027
Record Dates: First submitted 1999-11-01; First posted 2004-04-06 (Estimated); Last update posted 2014-09-10 (Estimated); Status verified 2014-09

CONDITIONS: Breast Cancer; Chronic Myeloproliferative Disorders; Gestational Trophoblastic Tumor; Kidney Cancer; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Neuroblastoma; Ovarian Cancer; Testicular Germ Cell Tumor
Keywords: stage IV breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; recurrent adult Hodgkin lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; refractory multiple myeloma; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; disseminated neuroblastoma; recurrent neuroblastoma; recurrent Wilms tumor and other childhood kidney tumors; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; chronic idiopathic myelofibrosis; testicular embryonal carcinoma; testicular choriocarcinoma; testicular teratoma; testicular yolk sac tumor; testicular embryonal carcinoma and teratoma; testicular embryonal carcinoma and teratoma with seminoma; testicular embryonal carcinoma and yolk sac tumor; testicular embryonal carcinoma and yolk sac tumor with seminoma; testicular embryonal carcinoma and seminoma; testicular yolk sac tumor and teratoma; testicular yolk sac tumor and teratoma with seminoma; testicular choriocarcinoma and yolk sac tumor; testicular choriocarcinoma and embryonal carcinoma; testicular choriocarcinoma and teratoma; testicular choriocarcinoma and seminoma; refractory hairy cell leukemia; recurrent ovarian germ cell tumor; ovarian yolk sac tumor; ovarian embryonal carcinoma; ovarian polyembryoma; ovarian choriocarcinoma; ovarian immature teratoma; ovarian mature teratoma; ovarian monodermal and highly specialized teratoma; ovarian mixed germ cell tumor; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; poor prognosis metastatic gestational trophoblastic tumor; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Breast Neoplasms; Myeloproliferative Disorders; Gestational Trophoblastic Disease; Kidney Neoplasms; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Neuroblastoma; Ovarian Neoplasms; Testicular Germ Cell Tumor; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Carcinoma, Ovarian Epithelial; Wilms Tumor; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Testicular Neoplasms; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Primary Myelofibrosis; Teratoma, Testicular; Endodermal Sinus Tumor; Teratoma; Seminoma; Carcinoma, Embryonal; Leukemia, Hairy Cell; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone | interventions — Interleukin-12 Subunit p35

INTERVENTIONS:
Biological: recombinant interleukin-12

SUMMARY:
RATIONALE: Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person's white blood cells to kill cancer cells.

PURPOSE: Phase I trial to study the effectiveness of interleukin-12 in treating patients who have hematologic cancer or solid tumor.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the safety and maximum tolerated dose of interleukin-12 (IL-12) in patients with hematologic malignancies or solid tumors who have undergone high-dose chemotherapy and autologous stem cell transplantation. II. Evaluate the hematologic and immunologic effects of IL-12 in these patients.

OUTLINE: This is a dose-escalation study. Patients receive interleukin-12 (IL-12) IV as a single test dose followed by 2 weeks of rest. Patients then receive IL-12 IV daily for 5 days followed by 16 days of rest for up to 6 courses. Cohorts of 3-5 patients receive escalating doses of IL-12 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 5 patients experience dose-limiting toxicity. Patients are followed until death.

PROJECTED ACCRUAL: A total of 12 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven hematologic malignancies or solid tumors Undergone high-dose chemotherapy or chemoradiotherapy with autologous bone marrow and/or peripheral blood stem cell transplantation Confirmation of complete remission is required for acute leukemia No significant CNS disease No clinically significant ascites or pleural effusions Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Not specified Menopausal status: Not specified Performance status: ECOG 0-1 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,000/mm3 Hemoglobin at least 9 g/dL (transfusion allowed) Platelet count at least 50,000/mm3 (transfusion independent) No clinically significant coagulopathy (unless due to cancer and resolved) Hepatic: Bilirubin no greater than 2 mg/dL SGOT no greater than 2 times upper limit of normal No chronic or acute hepatitis Hepatitis B surface antigen negative Renal: Creatinine no greater than 2 mg/dL No symptomatic hypercalcemia Calcium less than 12 mg/dL Cardiovascular: No uncontrolled angina No arrhythmias requiring drug or device therapy No symptomatic congestive heart failure Pulmonary: No clinically significant pulmonary dysfunction Metabolic: No uncontrolled diabetes mellitus No untreated hyper or hypothyroidism No Cushing's disease Gastrointestinal: No clinically significant gastrointestinal hemorrhages No uncontrolled peptic ulcer disease No history of inflammatory bowel disease Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No serious infection requiring IV antibiotics No psychosis No clinically significant autoimmune disease HIV negative

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics No concurrent biologic therapy Chemotherapy: See Disease Characteristics Endocrine therapy: At least 3 weeks since prior corticosteroids No concurrent systemic corticosteroids (other than replacement doses) Radiotherapy: See Disease Characteristics Surgery: Not specified Other: No other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1997-10

CONTACTS AND LOCATIONS:
Overall Officials: Michael J. Robertson, MD, Study Chair — Indiana University Melvin and Bren Simon Cancer Center
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States